CLINICAL TRIAL: NCT05944510
Title: Dextromethorphan as an Augmentation Agent in Treatment-resistant Schizophrenia: A Randomized, Group Sequential Adaptive Design, Controlled Clinical Trial
Brief Title: Dextromethorphan as an Augmentation Agent in Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMS BBSR/PGThesis/23-24/02
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Add-on Dextromethorphan (Experimental): Dextromethorphan 30mg once daily will be administered along with clozapine (as standard of care) in Treatment-resistant schizophrenia.
  Interventions: Drug: Dextromethorphan
- Add-on Placebo (Placebo Comparator): Matched Placebo will be administered along with clozapine (as standard of care) in Treatment resistant schizophrenia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — Dextromethorphan 30mg will be administered along with Clozapine (standard of care) in treatment resistant schizophrenia.
  Arms: Add-on Dextromethorphan
Drug: Placebo — Matched placebo will be administered along with Clozapine (standard of care) in treatment resistant schizophrenia.
  Arms: Add-on Placebo

SUMMARY:
Dextromethorphan acts as N-methyl-D-aspartate (NMDA) antagonist. In Treatment resistant schizophrenia(TRS) the efficacy of treatment response by clozapine is only around 40%. Numerous augmentation agent have been tried which includes antipsychotics, anticonvulsants, antidepressants and NMDA antagonist. The NMDA antagonist such as Riluzole and Memantine have shown good efficacy in TRS. Therefore we are evaluating NMDA antagonist, dextromethorphan in TRS. The dextromethorphan or placebo will be administered along with clozapine in TRS patients. The study is randomized double blind placebo controlled group sequential trial.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia patients who are diagnosed as treatment-resistant schizophrenia (TRS) defined as having been tried and not responded to any two antipsychotic medication for a duration of 6 weeks with dose equivalent of 600 mg of chlorpromazine and initiated on clozapine for the treatment of the same.
* The patients who are on stable dose of clozapine.
* Patients of either sex with age >18 years.
* Patients for whom legally authorized representative (LAR) are willing to give informed consent.

Exclusion Criteria:

* Patients with significant medical comorbidity.
* Patients with significant psychiatric comorbidity.
* Patients having active substance abuse history during the time of screening.
* Female patients who are pregnant or in reproductive age not using contraception.
* Female patients who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Positive and negative symptom scale score | Baseline and 12 weeks
  The change in symptom scoring of schizophrenia at 12 weeks from baseline using Positive and negative symptom scale in the study groups. On this scale, total minimum score= 30, maximum score= 210. Higher score denotes a worse outcome.

SECONDARY OUTCOMES:
Responder rate | 12 weeks
  To analyze and compare responder rate between study groups. The responder rate is defined as ≥ 20% reduction in PANSS score at 12 weeks from baseline.
Incidence of clozapine resistance | 12 weeks
  To evaluate the proportion of patients developing clozapine resistance after 12 weeks of therapy.
Requirement of clozapine dose modification | 12 weeks
  To evaluate the proportion of patients requiring clozapine dose increments or decrements over 12 weeks
Clinical global impression scoring | 12 weeks
  To evaluate for clinical status according to the clinical global impression scale. Clinical global impression is presented in a scale of 1-7. High score denotes a worse outcome.
Mini-mental state score | Baseline and 12 weeks
  The change in cognition as assessed by mini-mental state examination on a 30-point questionnaire at 12 weeks from baseline. Minimum and maximum score on this scale is 0 and 30. Lower score denotes worse outcome.
Serum clozapine level | Baseline and 12 weeks
  To evaluate serum clozapine levels (trough level) at baseline and follow-up at 12 weeks.
Incidence of treatment-emergent adverse events | 12 weeks
  To evaluate and compare the incidence of treatment-emergent adverse events in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, D.M., Study Chair — AIIMS Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No
Necessary data can be requested from the principal investigator.

REFERENCES:
- [Background] Siskind D, Siskind V, Kisely S. Clozapine Response Rates among People with Treatment-Resistant Schizophrenia: Data from a Systematic Review and Meta-Analysis. Can J Psychiatry. 2017 Nov;62(11):772-777. doi: 10.1177/0706743717718167. Epub 2017 Jun 28. PMID 28655284
- [Background] Vayisoglu S, Karahan S, Anil Yagcioglu AE. Augmentation of Antipsychotic Treatment with Memantine in Patients with Schizophrenia: A Systematic Review and Meta-Analysis. Turk Psikiyatri Derg. 2019 Winter;30(4):253-259. English, Turkish. PMID 32594486
- [Background] Kruse AO, Bustillo JR. Glutamatergic dysfunction in Schizophrenia. Transl Psychiatry. 2022 Dec 3;12(1):500. doi: 10.1038/s41398-022-02253-w. PMID 36463316
- [Background] de Boer JN, Vingerhoets C, Hirdes M, McAlonan GM, Amelsvoort TV, Zinkstok JR. Efficacy and tolerability of riluzole in psychiatric disorders: A systematic review and preliminary meta-analysis. Psychiatry Res. 2019 Aug;278:294-302. doi: 10.1016/j.psychres.2019.06.020. Epub 2019 Jun 21. PMID 31254879
- [Background] Siu A, Drachtman R. Dextromethorphan: a review of N-methyl-d-aspartate receptor antagonist in the management of pain. CNS Drug Rev. 2007 Spring;13(1):96-106. doi: 10.1111/j.1527-3458.2007.00006.x. PMID 17461892